CLINICAL TRIAL: NCT06296225
Title: Effect of Vibratory Tendon Stimulation on Muscle Fatigue in the Acute Post-stroke Phase : Vibramain1
Brief Title: Effect of Vibratory Tendon Stimulation on Muscle Fatigue in the Acute Post-stroke Phase
Acronym: VIBRAMAIN1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2023-07
Record Dates: First submitted 2024-02-12; First posted 2024-03-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Stroke, Acute; Fatigue
Keywords: Stroke; vibration; Handgrip strength; Fatigue
MeSH Terms: conditions — Stroke; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibration group (Experimental): Patients with acute stroke less than 7 days with only one paretic upper limb will be assessed for eligibility.
  Patient will undergo 8 grip strength evaluation and 30 minutes of forehand muscles vibration.
  Interventions: Device: Vibration

INTERVENTIONS:
Device: Vibration — Grip strenght measurement will always be done in the same way : for each series, 3 measurements of maximum strength will be taken for each side. Participants will receive verbal encouragement.
  After initial both sides grip strength evaluation, all participant will first experiment the vibration situation using the device Vibramoov Physio (TechnoConcept, Manosque, France): the vibrations had a frequency of 100Hz, with an amplitude of 2mm, they will be applied to the anterior part of the forearm for 10 minutes, 3 times. At the end of each 10 minutes vibration session, handgrip strength will be assessed.
  * Participants then have a one-hour rest period.
  * Control situation: participants will have 4 series of grip strength measurements every 10 minutes.
  At the end of the 2 hours, the patient will be discharged from the study protocol.
  Other Names: Handgrip Strength

SUMMARY:
It seems that prolonged vibratory stimulation of the anterior forearm in healthy subjects leads to fatigue of the muscles concerned, with a reduction in their strength. The aim of this study is to evaluate the impact of vibratory tendon stimulation on grip force fatigue during the acute post-stroke phase.

The investigations will be carried out by a specialized physiotherapist from the neurology department.

The experiment consists of three successive phases:

* First : measurement of the maximum handgrip force before any vibratory stimulation and then after the three sessions of ten-minute vibration.
* Second : Rest period
* Third: control phase with measurement of the maximum grip force every ten minutes without vibration.

ELIGIBILITY:
Inclusion Criteria:

* Age:18 to 85
* Acute stroke (less than 7 days)
* Paretic upper limb: 3 or 4 to the MRC score and able to obtain a value of at least 10 kilograms on the handgrip strength
* Able to sign a consent form
* Affiliated to a social insurance

Exclusion Criteria:

* Person under tutorship or curatorship,
* Sleepiness
* Pregnancy or breastfeeding woman

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Maximum handgrip strength measured by a digital dynamometer | 2 hours
  Handgrip strength in kilograms

SECONDARY OUTCOMES:
Fatigue evolution | 2 hours
  Fatigue assessed with Borg Scale : Minimal score indicates no fatigue (Minimum : 0 - Maximum : 10)
Evolution of handgrip strength during the vibration session measured by a digital dynamometer | 30 minutes
  Handgrip strength in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Canan OZSANCAK, MD, Study Chair — CHU ORLEANS
Locations (4):
- France (4):
  - CH de Chartres, Chartres
  - CHU d'ORLEANS, Orléans
  - Hopital Pitie Salpetriere, Paris
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Souron R, Besson T, Millet GY, Lapole T. Correction to: Acute and chronic neuromuscular adaptations to local vibration training. Eur J Appl Physiol. 2018 Feb;118(2):483. doi: 10.1007/s00421-017-3776-9. PMID 29218406
- [Background] Shirato R, Shimanuki R, Shoji T, Mugikura M. Inhibitory Effects of Prolonged Focal Muscle Vibration on Maximal Grip Strength and Muscle Activity of Wrist and Extrinsic Finger Flexor Muscles. J Chiropr Med. 2023 Jun;22(2):107-115. doi: 10.1016/j.jcm.2023.03.003. Epub 2023 Apr 21. PMID 37346243
- [Background] Toscano M, Celletti C, Vigano A, Altarocca A, Giuliani G, Jannini TB, Mastria G, Ruggiero M, Maestrini I, Vicenzini E, Altieri M, Camerota F, Di Piero V. Short-Term Effects of Focal Muscle Vibration on Motor Recovery After Acute Stroke: A Pilot Randomized Sham-Controlled Study. Front Neurol. 2019 Feb 19;10:115. doi: 10.3389/fneur.2019.00115. eCollection 2019. PMID 30873102
- [Background] Celletti C, Sinibaldi E, Pierelli F, Monari G, Camerota F. Focal Muscle Vibration and Progressive Modular Rebalancing with neurokinetic facilitations in post- stroke recovery of upper limb. Clin Ter. 2017 Jan-Feb;168(1):e33-e36. doi: 10.7417/CT.2017.1979. PMID 28240760
- [Background] Bobos P, Nazari G, Lu Z, MacDermid JC. Measurement Properties of the Hand Grip Strength Assessment: A Systematic Review With Meta-analysis. Arch Phys Med Rehabil. 2020 Mar;101(3):553-565. doi: 10.1016/j.apmr.2019.10.183. Epub 2019 Nov 13. PMID 31730754